CLINICAL TRIAL: NCT01912027
Title: Open Latarjet Techniques Versus Arthroscopic Latarjet Techniques on Anterior Shoulder Instability: The Comparison of Clinical and Radiographic Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fenglong Li, MD (Other)
Responsible Party: Sponsor-Investigator, Fenglong Li, MD, MD, Beijing Jishuitan Hospital
Organization: Beijing Jishuitan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JST1307A2; JST130701 (Other: Beijing Jishuitan Hospital)
Record Dates: First submitted 2013-07-18; First posted 2013-07-30 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Shoulder Instability

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arthroscopic Latarjet technique (Experimental): Arthroscopic Latarjet technique
  Interventions: Procedure: Arthroscopic Latarjet techniques
- Open Latarjet technique (Active Comparator): Open Latarjet technique
  Interventions: Procedure: Open Latarjet technique

INTERVENTIONS:
Procedure: Open Latarjet technique
  Arms: Open Latarjet technique
Procedure: Arthroscopic Latarjet techniques
  Arms: Arthroscopic Latarjet technique

SUMMARY:
The open Latarjet techniques has benn considered as an effective treatment on anterior shoulder instability.Over the past decade there has been a shift from open to all-arthroscopic technique in many surgeries. The arthroscopic technique may result in less postoperative stiffness and faster rehabilitation. So we hypothesized that the arthroscopic Latarjet techniques would have better clinical and radiographic outcomes than the open Latarjet Techniques on anterior shoulder instability.

ELIGIBILITY:
Inclusion Criteria:

* age older than 15 years
* Traumatic anterior shoulder instability
* Recurrent instability
* Glenoid defects larger than 25%
* Clinical and radiographic data at pre-operation and follow-up

Exclusion Criteria:

* Younger than 18 years
* Non-traumatic shoulder instability
* Primary episode of instability
* Glenoid defects less than 25%
* Previous surgical procedure Incomplete clinical or radiographic data Combination with rotator cuff tear

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
The functional and clinical outcomes are evaluated with the range of motion(ROM),VAS scores, UCLA scores, Constant scores, ASES scores and SST scores. The radiographic outcome is also assessed with X-ray plain film . | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Jiang, MD, Principal Investigator — Beijing Jishuitan Hospitial
Locations (2):
- China (2):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijng, Beijing Municipality